CLINICAL TRIAL: NCT02529839
Title: Safety and Efficacy of an Immunoablative Nonmyeloablative Conditioning Protocol for Autologous Bone Marrow Transplantation in Patients With Multiple Sclerosis
Brief Title: Safety and Efficacy of an Immunoablative Nonmyeloablative Conditioning Protocol for Autologous Bone Marrow Transplantation (BMT) in Patients With Multiple Sclerosis (MS)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0105-15-HMO-CTIL
Record Dates: First submitted 2015-06-10; First posted 2015-08-20 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-04

CONDITIONS: Multiple Sclerosis
Keywords: MS; BMT
MeSH Terms: conditions — Multiple Sclerosis | interventions — fludarabine; Cyclophosphamide; Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental (Experimental): Fludarabine 30mg/m2 for 4 days, Cyclophosphamide 50mg/kg for 2 days, Alemtuzumab administered subcutaneously 24mg total dose.
  Autologous bone marrow transplantation
  Interventions: Procedure: Autologous bone marrow transplantation; Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Alemtuzumab

INTERVENTIONS:
Procedure: Autologous bone marrow transplantation — IMMUNOABLATIVE NONMYELOABLATIVE AUTOLOGOUS BONE MARROW TRANSPLANTATION on Day 0
Drug: Fludarabine — 30mg/m2 on days -6 through -3
Drug: Cyclophosphamide — 50mg/kg on days -5 through -4
Drug: Alemtuzumab — 3mg on day -3, 9mg on day -2, 12 mg on day -1

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of an immunoablative nonmyeloablative conditioning protocol for autologous bone marrow transplantation in patients with Multiple Sclerosis. Patients meeting inclusion and exclusion criteria will start an immunoablative nonmyeloablative conditioning regimen followed by autologous bone marrow transplantation. Patients will be followed for one year by a neurologist to evaluate the course of the disease after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Consenting patients fulfilling the Poser's clinical criteria for definite MS
2. Age: 18-65, males and females
3. Relapsing and secondary progressive forms of MS with evidence of significant activity of MS (clinical and on the MRI).
4. EDSS score of 2.0 to 7.0 (see table 1).
5. Failure to at least one line of the currently available treatment, registered treatments (i.e. interferons, Copaxone, Tysabri, Gilenya, Tecfidera, immunosuppression) for MS. The lack of response to these treatments will be determined/defined by either an increase (deterioration) of one degree (or more) in the EDSS score, when baseline EDSS is less than 5.0 or 0.5 degree, when baseline EDSS is 5.0 or more, during the last year or the appearance of one major relapse of MS during the same period of time (under treatment), or evidence for new activity of MS (new T2 lesions or gadolinium enhancing lesions) during the last 12 months.
6. Duration of disease: >2 years, except cases with rapid progression, i.e. annual relapse rate ≥2 per 2 years on a conventional treatment or malignant multiple sclerosis with very intense symptoms (types is in most cases deadly).

Exclusion Criteria:

1. Patients suffering from significant cardiac, renal or hepatic failure or any other disease that may risk the patient or interfere with the ability to undergo high dose immunosuppression associated toxicities (according to the existing limitations for autologous transplantation).
2. Patients with active infections.
3. Patients with severe cognitive decline or inability to understand and sign the informed consent.
4. Patients who were treated with investigational protocols during the last 3 months prior to the inclusion.
5. Patients who received high dose immunosuppression with autologous stem cell rescue in the past with no effect.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Engraftment parameters of Neutrophils and Platelets | 1 year
  Absolute Neutrophil count >500 /microliter, Platelets>20,000/microliter
Transplant related mortality by Day 100 | Day 100

SECONDARY OUTCOMES:
Changes in the Expanded Disability Status Scale (EDSS score, as compared to baseline) | 1 year
Overall survival (OS) at 1 year | 1 year
Progression-free survival (PFS) at 1 year | 1 year
Changes in MRI activity | 1 year
  T2 number
Changes in MRI activity | 1 year
  Volume of gadolinium enhancing lesions

CONTACTS AND LOCATIONS:
Overall Officials: Igor Resnick, Prof., Principal Investigator — Bone Marrow Transplantation, Cancer Immunotherapy & Immunobiology Research Center, Hadassah University Hospital, Ein Kerem, Jerusalem, Israel